CLINICAL TRIAL: NCT00757458
Title: Evaluation of Bacterial and Fungal Contamination During Propofol Continuous Infusion in Patients Undergoing General Anesthesia
Brief Title: Evaluation of Bacterial and Fungal Contamination During Propofol Continuous Infusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Jose Otavio Costa Auler Jr. / Full Professor Department of Anesthesiology, Universidade de Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: EDTA-652
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Drug Contamination
Keywords: Propofol; Bacterial growth; Fungal growth; EDTA; Target controlled infusion
MeSH Terms: interventions — Edetic Acid; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): TCI with EDTA
  Interventions: Drug: EDTA without re-filling
- 2 (Active Comparator): Re-filling of propofol syringe (Diprivan®-Astra Zeneca) with propofol containing EDTA
  Interventions: Other: Propofol syringe re-filling with propofol containing EDTA
- 3 (Active Comparator): Re-filling of propofol syringe (Diprivan®-Astra Zeneca) with propofol without EDTA
  Interventions: Other: Re-filling of syringe with propofol without EDTA
- 4 (Active Comparator): Target controlled infusion of propofol without EDTA
  Interventions: Other: Target controlled infusion of propofol without EDTA

INTERVENTIONS:
Drug: EDTA without re-filling — Target controlled infusion of propofol containing EDTA (Diprivan®-Astra Zeneca) using equipment Diprifusor® (Astra Zeneca), without re-filling of syringe.
  Arms: 1
Other: Propofol syringe re-filling with propofol containing EDTA — Target controlled infusion of propofol (Diprivan®-Astra Zeneca) using equipment Diprifusor® (Astra Zeneca) with re-filling of syringe with propofol containing EDTA.
  Arms: 2
Other: Target controlled infusion of propofol without EDTA — Target controlled infusion of propofol without EDTA using Marshal´s technic with Alaris® or Fresenius® equipment
  Arms: 4
Other: Re-filling of syringe with propofol without EDTA — Target controlled infusion of propofol (Diprivan®-Astra Zeneca) using equipment Diprifusor® (Astra Zeneca) with re-filling of syringe with propofol not containing EDTA.
  Arms: 3

SUMMARY:
The purpose of this study is to verify the existence of bacterial and/or fungal contamination during different technics of propofol with or without EDTA continuous infusion in patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age eighteen years old or more
* ASA Physiological Status P1 ou P2
* Patients undergoing clean procedure under general anesthesia.

Exclusion Criteria:

* Patients under eighteen years old
* ASA Physiological Status P3, P4 or P5
* Current infectious process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Existence of bacterial and/or fungal contamination during different technics of propofol continuous infusion | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Sao Paulo Hospital das Clinicas, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Jansson JR, Fukada T, Ozaki M, Kimura S. Propofol EDTA and reduced incidence of infection. Anaesth Intensive Care. 2006 Jun;34(3):362-8. doi: 10.1177/0310057X0603400305. PMID 16802492
- [Background] Fukada T, Ozaki M. Microbial growth in propofol formulations with disodium edetate and the influence of venous access system dead space. Anaesthesia. 2007 Jun;62(6):575-80. doi: 10.1111/j.1365-2044.2007.05002.x. PMID 17506735
- [Background] Trepanier CA, Lessard MR. Propofol and the risk of transmission of infection. Can J Anaesth. 2003 Jun-Jul;50(6):533-7. doi: 10.1007/BF03018635. No abstract available. English, French. PMID 12826541
- [Background] Bennett SN, McNeil MM, Bland LA, Arduino MJ, Villarino ME, Perrotta DM, Burwen DR, Welbel SF, Pegues DA, Stroud L, et al. Postoperative infections traced to contamination of an intravenous anesthetic, propofol. N Engl J Med. 1995 Jul 20;333(3):147-54. doi: 10.1056/NEJM199507203330303. PMID 7791816